CLINICAL TRIAL: NCT01156168
Title: VEGF Gene Amplification/Deletion and Haplotype as Biomarkers for Bevacizumab in Breast Cancer
Brief Title: Biomarkers in Tissue Samples From Patients With Breast Cancer Treated With Bevacizumab
Status: Completed | Type: Observational
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Other Study IDs: CDR0000681004; ECOG-E2100T4
Record Dates: First submitted 2010-07-01; First posted 2010-07-02 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Breast Cancer
Keywords: male breast cancer; stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Gene Expression Profiling; Amplified Fragment Length Polymorphism Analysis; Immunohistochemistry

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

INTERVENTIONS:
Genetic: DNA analysis
Genetic: gene expression analysis
Genetic: polymorphism analysis
Genetic: protein expression analysis
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: DNA analysis of tumor tissue may help doctors predict how well patients will respond to treatment.

PURPOSE: This research study is studying biomarkers in tissue samples from patients with breast cancer treated with bevacizumab.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To demonstrate that vascular endothelial growth factor-A (VEGFA) haplotypes that are associated with an increased VEGFA expression will predict superior outcome for patients with metastatic breast cancer receiving bevacizumab in ECOG-E2100 (but not for the control arm).
* To demonstrate that candidate single nucleotide polymorphisms (SNPs) will further improve the predictive capacity of outcome (efficacy and toxicity) in patients enrolled in ECOG-E2100.
* To demonstrate that tumor VEGFA amplification or borderline amplification (estimated 14% frequency) will predict superior outcome for patients with metastatic breast cancer receiving bevacizumab on ECOG-E2100 whereas those with VEGFA deletion (estimated 11% frequency) will predict inferior outcome.
* To demonstrate that VEGFA amplification/deletion will not predict outcome in the control arm of ECOG-E2100.

Secondary

* To demonstrate that tumor VEGFA amplification will predict increased protein expression as ascertained by IHC.
* To demonstrate that a combined algorithm calculated from tumor-specific variability (VEGFA amplification/deletion) and host-specific variability (SNPs) will optimally predict outcome (efficacy) with bevacizumab in patients enrolled on ECOG-E2100.

OUTLINE: This is a multicenter study.

Previously collected tumor-derived DNA is analyzed for VEGFA amplification/deletion and haplotype as biomarkers for outcome after bevacizumab treatment. Gene expression, polymorphism, protein expression analysis, and IHC are performed on the samples.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Enrolled on ECOG-E2100

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Samples from patients enrolled on E2100 from whom samples were submitted for research
Sampling Method: Non-Probability Sample
Enrollment: 363 (Actual)
Dates: Start 2011-04-05 (Actual); Primary Completion 2011-09-08 (Actual); Study Completion 2011-09-08 (Actual)

PRIMARY OUTCOMES:
Comparison between VEGF haplotype and median overall survival (OS) and grade 3/4 hypertension (HTN) | 1 month

SECONDARY OUTCOMES:
Comparison between VEGF amplification/deletion and VEGF expression | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Bryan P. Schneider, MD, Principal Investigator — Indiana University Melvin and Bren Simon Cancer Center